CLINICAL TRIAL: NCT04148352
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dupilumab and Milk Oral Immunotherapy for the Treatment of Patients With Cow's Milk Allergy
Brief Title: Dupilumab and Milk OIT for the Treatment of Cow's Milk Allergy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Resources not available to continue study
Sponsor: Andrew J Long, PharmD (Other)
Collaborators: Robert Levin Charitable Fund (Unknown); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Andrew J Long, PharmD, Pharmacist, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-52976
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Allergies Food Milk
Keywords: Food allergy; Milk allergy; Oral Immunotherapy
MeSH Terms: conditions — Milk Hypersensitivity; Food Hypersensitivity | interventions — dupilumab

STUDY DESIGN:
Intervention Model Description: dupilumab or placebo arm
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (Experimental): 24-week treatment period, which includes a 4-week run-in period with dupilumab followed by 12 weeks of treatment with dupilumab in combination with a gradual up-dosing of milk protein OIT, then followed by 8 weeks of milk OIT dosing with no dupilumab
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): 24-week treatment period, which includes a 4-week run-in period with placebo for dupilumab followed by 12 weeks of treatment with placebo for dupilumab in combination with a gradual up-dosing of milk protein OIT, then followed by 8 weeks of milk OIT dosing with no placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab — Dupilumab injected every 2 weeks for 18 weeks
  Arms: Dupilumab
Other: Placebo — Placebo injected every 2 weeks for 18 weeks
  Arms: Placebo

SUMMARY:
This is a phase 2, multicenter, randomized, double-blind, parallel group, 2 arm study in approximately 40 subjects aged 4 to 50 years, inclusive, who are allergic to cow's milk. The primary objective is to assess whether dupilumab as an adjunct to milk oral immunotherapy (OIT) compared to placebo improves the safety of milk OIT and rates of desensitization, defined as an increase in the proportion of subjects who pass a double-blind placebo-controlled food challenge (DBPCFC) to at least 2040 mg cumulative milk protein at week 18.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 50 years (inclusive)
* Clinical history of allergy to cow's milk or milk-containing foods
* Serum IgE to milk of >4 kUA/L within the last 12 months and/or a SPT to milk ≥6 mm compared to a negative control
* Experience clinical reaction at or before 444 mg cumulative protein dose of cow's milk protein on Screening DBPCFC
* No clinical reaction observed during the placebo (oat) Screening DBPCFC
* Subjects with other known food allergies must agree to eliminate these other food items from their diet so as not to confound the safety and efficacy data from the study
* Use of effective birth control by female participants of childbearing potential

Exclusion Criteria:

* Any previous exposure to dupilumab
* Known hypersensitivity to dupilumab or any of its excipients
* Known hypersensitivity to epinephrine or any of its excipients
* Allergy to oat (placebo in DBPCFC)
* History of severe anaphylaxis to cow's milk, defined as neurological compromise or requiring intubation
* Recent history of frequent severe, life-threatening episodes of anaphylaxis or anaphylactic shock as defined as 3 or more episodes of anaphylaxis within the past year
* Inability to tolerate biological (antibody) therapies
* Body weight <5 kg at the time of screening
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia (e.g., difficulty swallowing, food "getting stuck"), or recurrent gastrointestinal symptoms of undiagnosed etiology
* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* History of a mast cell disorder
* Established diagnosis of a primary immunodeficiency disorder
* Severe asthma or mild or moderate asthma if uncontrolled or difficult to control
* Current participation or within the last 4 months in any other interventional study
* Use of medication such as beta-blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Pregnant or breastfeeding women

Ages: 4 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Long, PharmD, Study Director — Stanford, Sean N. Parker Center for Allergy & Asthma Research
Locations (3):
- United States (3):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Sean N. Parker Center for Allergy & Asthma Research at Stanford University, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghelli C, Costanzo G, Canonica GW, Heffler E, Paoletti G. New evidence in food allergies treatment. Curr Opin Allergy Clin Immunol. 2024 Aug 1;24(4):251-256. doi: 10.1097/ACI.0000000000000999. Epub 2024 May 30. PMID 38814736

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 33 enrolled, 8 participants failed at screening and 2 withdrew from the study prior to randomization, for a total of 10 participants consented but not randomized
Groups:
- Active Dupilumab and Milk Oral Immunotherapy (OIT): Dupilumab every two to four weeks for 4 weeks, followed by dupilumab every two to four weeks plus milk OIT for 12 weeks, then milk OIT alone for 8 weeks
- Placebo for Dupilumab and Milk OIT: Placebo for dupilumab every two to four weeks for 4 weeks, followed by placebo for dupilumab every two to four weeks plus milk OIT for 12 weeks, then milk OIT alone for 8 weeks
Period: Overall Study
Arm/Group | Active Dupilumab and Milk Oral Immunotherapy (OIT) | Placebo for Dupilumab and Milk OIT
Started | 11 | 12
Week 18 Double-Blind, Placebo-Controlled Food Challenge (DBPCFC) | 11 | 8
Week 24 DBPCFC | 11 | 6
Completed | 11 | 6
Not Completed | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Active Dupilumab and Milk OIT: Dupilumab every two to four weeks for 4 weeks, followed by dupilumab every two to four weeks plus milk OIT for 12 weeks, then milk OIT alone for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Customized [Count of Participants; unit: Participants]
  4 - 10 years | 4 | 6 | 10
  11 - 17 years | 4 | 3 | 7
  18+ years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 5 | 12
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
History of Atopy [Count of Participants; unit: Participants]
  Asthma | 7 | 8 | 15
  Allergic Rhinitis | 6 | 6 | 12
  Atopic Disease | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Treated With Dupilumab Plus Milk Protein OIT vs Placebo Plus Milk Protein OIT Who Tolerate at Least 2040 mg (Cumulative) Cow's Milk Protein During DBPCFC to Milk at Week 18
Description: DBPCFC double-blind, placebo-controlled food challenge; OIT oral immunotherapy; withdrawals are imputed as failures
Time Frame: Week 18
Population: Intention to treat population: all randomized patients, analyzed in the treatment group they were assigned to, regardless of whether they actually received the treatment, dropped out, or deviated from the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 8 | 5

2. Secondary Outcome: Proportion of Participants Who Tolerate at Least 1040 mg Cumulative Milk Protein at Week 18 DBPCFC
Description: DBPCFC double-blind, placebo-controlled food challenge; withdrawals are imputed as failures
Time Frame: Week 18
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 9 | 6

3. Secondary Outcome: Proportion of Participants Who Tolerate 4040 mg Cumulative Milk Protein at Week 18 DBPCFC
Description: DBPCFC double-blind, placebo-controlled food challenge; withdrawals are imputed as failures
Time Frame: Week 18
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 5 | 3

4. Secondary Outcome: Proportion of Participants Who Tolerate at Least 1040 mg Cumulative Milk Protein at Week 24 DBPCFC
Description: DBPCFC double-blind, placebo-controlled food challenge; withdrawals are imputed as failures
Time Frame: week 24
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 8 | 5

5. Secondary Outcome: Proportion of Participants Who Tolerate at Least 2040 mg Cumulative Milk Protein at Week 24 DBPCFC
Description: DBPCFC double-blind, placebo-controlled food challenge; withdrawals are imputed as failures
Time Frame: Week 24
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 7 | 5

6. Secondary Outcome: Proportion of Participants Who Tolerate 4040 mg Cumulative Milk Protein at Week 24 DBPCFC
Description: DBPCFC double-blind, placebo-controlled food challenge; withdrawals are imputed as failures
Time Frame: Week 24
Population: Intention to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 12
Participants | 5 | 3

7. Secondary Outcome: Change in the Cumulative Tolerated Dose (CTD) of Milk Protein During DBPCFC From Baseline to Week 18 Across Cohorts as Pairwise Comparisons of All Treatment Groups
Description: Baseline values reflect the log10 of cumulative tolerated dose (CTD) of milk protein. The change metric reflects the order of magnitude of paired differences in CTD between baseline and week 18.
Time Frame: Baseline and week 18
Population: Participants with week 18 data
Measure: Mean (Standard Deviation); unit: log10 mg cumulative tolerated protein
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 8
log10 mg cumulative tolerated protein
  Baseline | 1.632 (0.888) | 1.899 (0.600)
  Change at week 18 | 1.574 (0.880) | 1.127 (0.618)

8. Secondary Outcome: Change in the Cumulative Tolerated Dose (CTD) of Milk Protein During DBPCFC From Baseline to Week 24 Across Cohorts as Pairwise Comparisons of All Treatment Groups
Description: Baseline values reflect the log10 of cumulative tolerated dose (CTD) of milk protein. The change metric reflects the order of magnitude of paired differences in CTD between baseline and week 24.
Time Frame: Baseline and week 24
Population: Participants with week 24 data
Measure: Mean (Standard Deviation); unit: log10 mg cumulative tolerated protein
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
Number analyzed (Participants) | 11 | 6
log10 mg cumulative tolerated protein
  Baseline | 1.632 (0.888) | 1.898 (0.691)
  Change at week 24 | 1.559 (1.153) | 1.366 (0.490)

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 24 weeks
Groups:
- Placebo for Dupilumab and Milk OIT: Dupilumab every two to four weeks for 4 weeks, followed by dupilumab every two to four weeks plus milk OIT for 12 weeks, then milk OIT alone for 8 weeks
Arm/Group | Active Dupilumab and Milk OIT | Placebo for Dupilumab and Milk OIT
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 10/11 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Dupilumab and Milk OIT (N=11) | Placebo for Dupilumab and Milk OIT (N=12)
Gastrointestinal Allergic AEs related to OIT (Gastrointestinal disorders) | 10 | 11
Skin Allergic AEs related to OIT (Skin and subcutaneous tissue disorders) | 8 | 9
Respiratory Allergic AEs related to OIT (Respiratory, thoracic and mediastinal disorders) | 6 | 10
General Allergic AEs related to OIT (General disorders) | 4 | 3
Nervous system Allergic AEs related to OIT (Nervous system disorders) | 1 | 1
Eye Allergic AEs related to OIT (Eye disorders) | 2 | 1
Immune system Allergic AEs related to OIT (Immune system disorders) | 1 | 2
Vascular Allergic AEs related to OIT (Vascular disorders) | 1 | 1
Gastrointestinal Food Challenge Reactions Allergic not related to OIT (Gastrointestinal disorders) | 7 | 7
Skin Food Challenge Reactions Allergic not related to OIT (Skin and subcutaneous tissue disorders) | 6 | 9
Respiratory Food Challenge Reactions Allergic not related to OIT (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Nervous System Food Challenge Reactions Allergic not related to OIT (Nervous system disorders) | 1 | 3
Psychiatric Food Challenge Reactions Allergic not related to OIT (Psychiatric disorders) | 2 | 0
Eye Food Challenge Reactions Allergic not related to OIT (Eye disorders) | 1 | 0
Immune System Food Challenge Reactions Allergic not related to OIT (Immune system disorders) | 1 | 2
General/administration site Non-Allergic not related to OIT (General disorders) | 4 | 3
Eye Non-Allergic not related to OIT (Eye disorders) | 1 | 0
Gastrointestinal Non-Allergic not related to OIT (Gastrointestinal disorders) | 2 | 1
Infection Non-Allergic not related to OIT (Infections and infestations) | 3 | 4
Nervous Non-Allergic not related to OIT (Nervous system disorders) | 3 | 1
Respiratory Non-Allergic not related to OIT (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Skin Non-Allergic not related to OIT (Skin and subcutaneous tissue disorders) | 0 | 2
Renal/Urinary Non-Allergic not related to OIT (Renal and urinary disorders) | 1 | 0
Injury Non-Allergic not related to OIT (Injury, poisoning and procedural complications) | 0 | 1
Ear Non-Allergic not related to OIT (Ear and labyrinth disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study findings are limited by the small sample size and high attrition. Screen failures and early loss to follow-up reduced power and may limit the ability to draw definitive conclusions about the intervention's effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT04148352/Prot_SAP_000.pdf